CLINICAL TRIAL: NCT03832582
Title: Prognostic of Annexin Imaging in Dissection of the Descending Aorta
Brief Title: Annexin Imaging in Dissection of the Descending Aorta
Acronym: PAIDDA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P1700905J
Record Dates: First submitted 2018-09-10; First posted 2019-02-06 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2018-09

CONDITIONS: Chronic Dissection of Thoracic Aorta (Disorder)
Keywords: Aorta; Type B dissection; Descending aorta dissection; Annexin
MeSH Terms: conditions — Dissection, Thoracic Aorta | interventions — Annexins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Annexin (Experimental): All patients will undergo a 99mTc-annexin V-128 scintigraphy (SPECT)
  Interventions: Drug: Annexin

INTERVENTIONS:
Drug: Annexin — All patients will undergo a 99mTc-annexin V-128 scintigraphy (SPECT)
  Other Names: Annexin scintigraphy

SUMMARY:
The relationship between the presence of a partial thrombus and aortic dilation after type B dissection has recently been reported. The originality lies in the idea of imaging thrombus activity to predict dilation after type B dissection. The innovative character is based on the use of annexin scintigraphy.

DETAILED DESCRIPTION:
To establish the proof of concept in humans of the link between the intensity of 99mTc-annexin V-128 binding in the descending thoracic aorta and the progression of aortic diameter in patients with type B aortic dissection.

ELIGIBILITY:
Inclusion Criteria:

* patient whose age is ≥ 18 years old
* any patient seen more than 6 months and less than 5 years after a dissection involving the descending aorta at Bichat Hospital, whether it is a dissection of the descending aorta alone or a dissection of the ascending aorta extended to the descending aorta
* dissection of the uncomplicated descending thoracic aorta: not requiring surgery or stent implantation within the first 6 months after acute dissection
* effective contraception for women of childbearing age

Exclusion Criteria:

* scheduled procedure for dissection of the descending aorta
* contraindication to aortic CT with injection of contrast media: renal failure with creatinine clearance <30 ml/min or creatinine >200 µmol/l; allergy to contrast media
* history of surgery or stent implantation in the descending thoracic aorta
* pregnant or breastfeeding women
* patient under guardianship or trusteeship
* non affiliation to social security or CMU (beneficiary or assignee)
* patient refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between the rate of expansion of the aortic diameter and the intensity of attachment of the annexin by the aortic wall descending | 30 months
  Pearson correlation coefficient between the rate of expansion of the aortic diameter measured by CT (at 6 months, 18 months and 30 months) in mm/year (at the site of maximum expansion) and the intensity of attachment of the annexin by the aortic wall descending in scintigraphy.

SECONDARY OUTCOMES:
Determination of the optimal threshold for annexin fixation to predict the evolution of aortic dilation (< 2 mm/year, >=2mm year) using ROC curve. | 30 months
  Determination of the optimal threshold for annexin fixation to predict the evolution of aortic dilation (< 2 mm/year, >=2mm year) using ROC curve. The cut-off point will be defined by the Youden index.
Blood level of fibrinolysis markers (D dimers, plasmin/anti-plasmin complexes) | 30 months
  Blood level of fibrinolysis markers (D dimers, plasmin/anti-plasmin complexes)
Blood level of thrombus procoagulant activity markers (circulating P-selectin and thrombin/anti-thrombin complexes) | 30 months
  Blood level of thrombus procoagulant activity markers (circulating P-selectin and thrombin/anti-thrombin complexes)
Morphological characteristics of the wall thrombus | 30 months
  Morphological characteristics of the wall thrombus: no thrombus of the false lumen, partial thrombosis or total thrombosis of the false lumen.
Determination of potential predictive clinical factors of aortic dilation rate | 30 months
  Determination of potential predictive clinical factors of aortic dilation rate: age, blood pressure, heart rate, sex, history of dissection, etiology (Marfan or no Marfan)
Determination of potential predictive SPECT factors of aortic dilation rate | 30 months
  Determination of potential predictive SPECT factors of aortic dilation rate: anormal annexin binding, ratio of annexin binding (TBR = Target-to-Background Ratio)
Determination of potential predictive biological factors of aortic dilation rate | 30 months
  Determination of potential predictive biological factors (C-Reactive Protein) of aortic dilation rate
Determination of potential predictive morphological factors of aortic dilation rate | 30 months
  Determination of potential predictive morphological factors of aortic dilation rate: no thrombus, partial thrombosis or total thrombosis.
Number of cardiovascular events | 30 months
  Number of cardiovascular events: cardiovascular death, dissection complications (including aortic rupture, malperfusion, emboli), aortic surgery.
Evaluation of the tolerance of the annexin scintigraphy by collecting side effects occurence | 3 days
  Tolerance of the annexin scintigraphy will be assessed using a questionnaire during a phone call at day 3 to ask the patients about side effects occurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Milleron, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Cardiologie - Hôpital Bichat Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided